CLINICAL TRIAL: NCT02778230
Title: Efficacy of Pea Hull Fibre Supplementation on Gastrointestinal Transit Time-induced Reduction in Proteolytic Fermentation and Enhancement of Wellness in Older Adults.
Brief Title: Efficacy of Pea Hull Fibre Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Saskatchewan Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201600646
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: fiber; gastrointestinal; microbiota

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pea Fiber (Experimental): Two fiber snacks fortified with 5 g/each of pea fiber (Best Pea Fiber 200) will be consumed each day for a period of two weeks.
  Interventions: Dietary Supplement: Pea Fiber
- Control (Other): Two control snacks will be consumed each day for a period of two weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Pea Fiber — Snacks (2 baked goods) fortified with 5 g pea hull fiber
  Arms: Pea Fiber
Dietary Supplement: Control — Snacks (2 baked goods) without fiber fortification.
  Arms: Control

SUMMARY:
The purpose of this randomized, cross-over study is to explore the effects of pea hull fiber on bowel movement frequency, transit time, appetite, gastrointestinal symptoms, microbiota composition and activity.

DETAILED DESCRIPTION:
A 10-week randomized, cross-over study will be carried out to assess the efficacy of pea hull fiber. Participants will complete a 2-week baseline period during which appetite, gastrointestinal symptoms, stool frequency, and stool consistency (transit time) will be collected by paper questionnaire, and participants will collect a single stool. Dietary data (24-hour dietary recalls) will be obtained via phone interviews 3 times during the baseline period. On or about day 15, participants will attend a study visit and complete the Simplified Nutritional Appetite Questionnaire (SNAQ) and Gastrointestinal Symptom Response Scale (GSRS). Participants will be randomized on or about day 15 and consume snacks without pea hull fiber for a 2-week control period, and snacks with added pea hull fiber for a 2-week treatment period separated by a 2-week washout period. In both intervention periods, participants will complete daily questionnaires to assess appetite, gastrointestinal symptoms, and stool frequency and consistency (transit time). Furthermore, they will complete SNAQ and GSRS after the end of each intervention period. The 24-hour dietary recalls will also be collected 3 times during each of the intervention periods. Participants will undergo an additional 2-week washout period after the second intervention period. During washout periods, the same data will be collected as was done during the baseline and intervention periods.Participants will be asked to collect one stool during pre-baseline and weeks 4, 6, 8 and 10 for a total of 5 stools. Stool samples will be analyzed for changes in the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Willing to have height and weight measured and provide demographic information (e.g. age, race, sex).
* Willing to consume pea hull fiber and control snacks daily each for a 2-week period
* Willing to complete a daily questionnaire regarding general and gastrointestinal wellness throughout the entire 10-weeks study.
* Willing to complete the GSRS (Gastrointestinal Symptom Rating Scale) and SNAQ questionnaires bi-weekly at study appointments.
* Willing to be interviewed for a 24-hr food recall, 3 times per 2-weeks period throughout the study.
* Willing to provide 5 stool samples, one in each 2-weeks period throughout the study.
* Willing and be able to provide a valid social security for study payment purposes.

Exclusion Criteria:

* Have any known food allergies.
* Are currently taking medications for diarrhea.
* Have taken antibiotics within the past four weeks prior to randomization.
* Are currently taking probiotics supplements and do not want to discontinue a minimum of two weeks prior to the study.
* Have previously or are currently being treated for any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's, Celiac, ulcerative colitis, etc.).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Stool consistency rating by Bristol Stool Form Scale | Changes from baseline to week 4, 6, 8 and 10.
  Assesses estimated transit time.

SECONDARY OUTCOMES:
Number of bowel movements per day averaged by week | Changes from baseline to week 4, 6, 8, and 10
  stool frequency
Microbiota profile changes: percent change at phylum and genus levels; changes in OTUs | Changes from baseline to week 4, 6, 8, and 10
GSRS (Gastrointestinal Symptom Response Scale) score. | Changes from baseline to week 4, 6, 8, and 10
SNAQ (Simplified Nutritional Appetite Questionnaire) score. | Changes from baseline to week 4, 6, 8, and 10

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Department, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
No current plan.

REFERENCES:
- [Derived] Alyousif Z, Mendoza DR, Auger J, De Carvalho V, Amos S, Sims C, Dahl WJ. Gastrointestinal Tolerance and Microbiome Response to Snacks Fortified with Pea Hull Fiber: A Randomized Trial in Older Adults. Curr Dev Nutr. 2020 Jan 17;4(2):nzaa005. doi: 10.1093/cdn/nzaa005. eCollection 2020 Feb. PMID 32025615